CLINICAL TRIAL: NCT01762891
Title: CI(R)CA : Coumadin Interaction With Rofecoxib, Celecoxib and Acetaminophen. A Prospective Double-blind, Placebo Controlled Study.
Brief Title: CI(R)CA : Coumadin Interaction With Rofecoxib, Celecoxib and Acetaminophen
Acronym: CI(R)CA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario Pedro Ernesto (Other)
Responsible Party: Principal Investigator, Veronica Silva Vilela, Physician, Hospital Universitario Pedro Ernesto
Allocation: Not Applicable | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 32323232; Pfizer (Other Grant/Funding Number: Pharmaceutic company)
Record Dates: First submitted 2009-09-24; First posted 2013-01-08 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2013-01

CONDITIONS: Antiphospholipid Antibody Syndrome
Keywords: Coumadin; celecoxib; rofecoxib; acetaminophen; antiphospholipid syndrome and INR
MeSH Terms: conditions — Antiphospholipid Syndrome | interventions — Celecoxib; Acetaminophen; rofecoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Celecoxib (Experimental): Celecoxib 200mg/day oral rout Intervention: celecoxib 200mg oral rout administered durng 15 days and followed by administration of rofecoxib 25mg/day during 15 days, placebo 15 days and acetaminophen 3g/day during 15 days.
  Interventions: Drug: Celecoxib; Drug: Acetaminophen; Drug: Rofecoxib; Drug: placebo

INTERVENTIONS:
Drug: Celecoxib — celecoxib 200mg/day by oral rout during 15 days followed by the administration of rofecoxib 25mg/day, acetaminophen 3g/day and placebo during 15 days each drug.
  Other Names: celebrex
Drug: Acetaminophen — Acetaminophen 3g/ was given during 15 days by oral rout following one of the other interventions or as the final intervention.
  Other Names: Tylenol
Drug: Rofecoxib — Rofecoxib 25mg/day was given by oral rout during 15 days following one or more interventions or as the final intervention.
  Other Names: Vioxx
Drug: placebo — Placebo pills were given during 15 days by oral rout as one of the four interventions.

SUMMARY:
Coumadin drug-drug interactions (DDI) are frequent. Patients in permanent use of coumadin are advised to avoid traditional nonsteroidal antiinflammatory drugs to avoid risk of bleeding. New selctive cyclooxygesase 2 inhibitors arisen as potential option for treating pain and inflamation in these patients once interactions with coumadin are supposed to be lower. The CI(R)CA study was made to evaluate in a prospective fashion the occurrence of DDI with new cyclooxygenase antiinflammatory drugs and coumadin when compared to acetaminophen and placebo.

DETAILED DESCRIPTION:
The CI(R)CA study included patient diagnosed with antiphospholipid syndrome in permanent use of coumadin. Eligible patients were invited to use in a prospective cross-over mode two weeks of celecoxib, rofecoxib, acetaminophen and placebo with two weeks of wash out between drugs. Their international normalized ratio (INR) were measured before and during the use of each study drug. The interaction with coumadin was evaluated according to increases or decreases on the INR after each medication.

ELIGIBILITY:
Inclusion Criteria:

* PAPS on contious stable dose of coumadin
* 18 years old or older
* Younger than 65 yo
* Signed informed consent.

Exclusion Criteria:

* Renal failure
* Heart failure
* Symptomatic gastritis or peptic ulcer
* Elevated liver enzymes (>3 fold)
* Platelet count < 100,000.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2003-03; Primary Completion 2006-07 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
International Normalized Ratio | increase or decrease on the INR after coxibs or placebo use during 15 days
  The outcome measure was verified 15 days after each intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Veronica S Vilela, MD, Principal Investigator — Hospital Universitario Pedro Ernesto